CLINICAL TRIAL: NCT02144675
Title: A Randomized Phase II Study of Nuclear Factor-kappa B (NF-κB) Inhibition During Induction Chemotherapy for Patients With Acute Myelogenous Leukemia
Brief Title: Choline Magnesium Trisalicylate and Combination Chemotherapy in Treating Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Rutgers Cancer Institute of New Jersey (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Roger Strair, MD, PhD, Professor of Medicine, RWJMS, Rutgers Cancer Institute of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0220080282; NCI-2012-00516 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0220080282 (Other: IRB number); P30CA072720 (NIH); 020803 (Other: Rutgers Cancer Institute of New Jersey)
Record Dates: First submitted 2014-05-20; First posted 2014-05-22 (Estimated); Results first posted 2018-07-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Recurrent Adult Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — choline magnesium trisalicylate; Idarubicin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (choline magnesium trisalicylate and chemotherapy) (Experimental): Patients receive choline magnesium trisalicylate PO every 8 hours on days 0-7, idarubicin IV on days 1-3, and cytarabine IV continuously on days 1-7.
  Interventions: Drug: choline magnesium trisalicylate; Drug: idarubicin; Drug: cytarabine; Other: laboratory biomarker analysis
- Arm II (chemotherapy) (Active Comparator): Patients receive idarubicin IV on days 1- 3 and cytarabine IV continuously on days 1-7.
  Interventions: Drug: idarubicin; Drug: cytarabine; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: choline magnesium trisalicylate — Given PO
  Other Names: Trilisate; Trisalicylate
  Arms: Arm I (choline magnesium trisalicylate and chemotherapy)
Drug: idarubicin — Given IV
  Other Names: 4-demethoxydaunorubicin; 4-DMDR; DMDR; IDA
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase II trial studies how well choline magnesium trisalicylate with idarubicin and cytarabine works in treating patients with acute myeloid leukemia. Drugs used in chemotherapy, such as choline magnesium trisalicylate, idarubicin, and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. It is not yet know whether choline magnesium trisalicylate and combination chemotherapy is more effective than combination chemotherapy alone in treating patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine temporal changes in leukemic cell nuclear factor of kappa light chain enhancer of B-cells 1 (NF-kB) activity when salicylate (choline magnesium trisalicylate) is administered to patients with acute myeloid leukemia (AML) during induction chemotherapy.

II. To determine toxicities associated with administration of salicylate in the setting of induction chemotherapy.

III. To determine if salicylate alters the expression of NF-kB-regulated genes in AML cells.

IV. To determine if NF-kB modulation by salicylate alters AML chemotherapy drug efflux.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive choline magnesium trisalicylate orally (PO) every 8 hours on days 0-7, idarubicin intravenously (IV) on days 1-3, and cytarabine IV continuously on days 1-7.

ARM II: Patients receive idarubicin IV on days 1-3 and cytarabine IV continuously on days 1-7.

In both arms, treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of non-M3 AML (patients with M3 subtype are excluded); determination of the presence of cytogenetic abnormalities will be by standard cytogenetics +/- fluorescent-in-situ (FISH) studies; additional molecular analyses for nucleophosmin (NPM) mutation and fms-related tyrosine kinase 3 (flt3) internal tandem duplication will be obtained as a part of standard care by institutional procedures
* Leukemic blast count > 1500/mm^3 of peripheral blood
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status =< 3
* Total bilirubin < 2 times the institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) < 3 times the institutional ULN
* Serum creatinine < 1.5 times the institutional ULN
* Multi gated acquisition scan (MUGA) or echocardiogram with left ventricular ejection fraction (LVEF) > 50%
* Women of childbearing potential must have a negative pregnancy test
* No uncontrolled psychiatric illness that the principal investigator feels will compromise obtaining informed consent from a patient
* Patient must be informed of the investigational nature of this study and must give written informed consent in accordance with institutional and federal guidelines; patients who do not provide informed consent will not be eligible for the study

Exclusion Criteria:

* Any coexisting medical condition or medications precluding full compliance with any of the arms of the study
* Allergies to any investigational drugs and/or to the chemotherapeutic agents
* Allergies to any non-steroidal anti-inflammatory drugs (NSAIDs)/salicylates (e.g., aspirin)
* Endoscopically documented upper or lower gastrointestinal (GI) related hemorrhage within last 6 months; also, patients with a clinical diagnosis of GI bleeding requiring blood transfusions will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-01; Primary Completion 2016-04-26 (Actual); Study Completion 2016-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Strair, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited through the Rutgers Cancer Institute of New Jersey. The study was open to accrual on 10/31/2008 and completed on 01/06/2015. All participants visits were completed and the study was closed by the Principal Investigator on 04/26/2016.
Period: Overall Study
Arm/Group | Arm I (Choline Magnesium Trisalicylate and Chemotherapy) | Arm II (Chemotherapy)
Started | 13 | 14
Completed | 13 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Choline Magnesium Trisalicylate and Chemotherapy) | Arm II (Chemotherapy) | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 19
  >=65 years | 3 | 5 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 7 | 4 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 12 | 14 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 11 | 13 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Inhibition of NF-kB Target Transcripts and/or Inhibition of Drug Efflux in at Least 50% of Patients
Description: The clinical trial will be based on a sequential monitoring so that we will have a 90% confidence that choline magnesium trisalicylate (CMT) based modulation of NF-kB transcriptional targets and/or drug efflux occurs in at least 50% of patients.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Choline Magnesium Trisalicylate and Chemotherapy) | Arm II (Chemotherapy)
Number analyzed (Participants) | 13 | 14
Participants | 13 | 14
Statistical Analysis 1: Comparison: Arm I (Choline Magnesium Trisalicylate and Chemotherapy) vs Arm II (Chemotherapy); Test type: Other; p < .05, Regression, Cox

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of approximately 1.5 months.
Arm/Group | Arm I (Choline Magnesium Trisalicylate and Chemotherapy) | Arm II (Chemotherapy)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 1/13 | 0/14
Other Adverse Events (participants affected / at risk) | 7/13 | 10/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Choline Magnesium Trisalicylate and Chemotherapy) (N=13) | Arm II (Chemotherapy) (N=14)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Choline Magnesium Trisalicylate and Chemotherapy) (N=13) | Arm II (Chemotherapy) (N=14)
Alkalosis (metabolic or respiratory) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Dermal change lymphedema, phlebolymphedema (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1) | 0 (0)
Low Platelets (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infe (Infections and infestations) | 1 (1) | 4 (4)
Low Hemoglobin (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils - Lung (pneumonia) (Infections and infestations) | 1 (1) | 0 (0)
Glucose, serum-high (hyperglycemia) (General disorders) | 1 (1) | 0 (0)
Potassium, serum-low (hypokalemia) (General disorders) | 1 (1) | 0 (0)
Calcium, serum-low (hypocalcemia) (General disorders) | 1 (1) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 0 (0) | 1 (1)
Heartburn/dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (inflammation of the small bowel) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pain - Abdomen NOS (General disorders) | 0 (0) | 1 (1)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 0 (0) | 2 (2)
Pain - Head/headache (General disorders) | 0 (0) | 1 (1)
Pain - Sore Throat (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No